CLINICAL TRIAL: NCT02254005
Title: An Open Phase I Single Dose Escalation Study of Bivatuzumab Mertansine Administered Intravenously in Female Patients With CD44v6 Positive Metastatic Breast Cancer With Repeated Administration in Patients With Clinical Benefit
Brief Title: Single Dose Escalation Study of Bivatuzumab Mertansine in Female Patients With CD44v6 Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1191.1
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — bivatuzumab mertansine

ARMS (1):
- single dose escalation (Experimental)
  Interventions: Drug: bivatuzumab mertansine

INTERVENTIONS:
Drug: bivatuzumab mertansine

SUMMARY:
Maximum tolerated dose (MTD), safety, pharmacokinetics, efficacy of bivatuzumab mertansine

ELIGIBILITY:
Inclusion Criteria:

1. female patients aged 18 years or older
2. patients with breast cancer positive for CD44v6 in at least 50 % of the tumour cells
3. patients with metastases pretreated with anthracyclines and taxanes (unless contraindications to taxanes and / or anthracyclines) or not amenable to established treatments
4. measurable tumour deposits by one or more radiological techniques (MRI, CT)
5. life expectancy of at least 6 months
6. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
7. patients must have given written informed consent (which must be consistent with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation)

Exclusion Criteria:

1. hypersensitivity to humanised or murine antibodies, immunoconjugates or the excipients of the trial drugs
2. known secondary malignancy requiring therapy
3. active infectious disease
4. brain metastases requiring therapy
5. neuropathy common toxicity criteria (CTC) grade 2 or above
6. absolute neutrophil count less than 1,500/mm3
7. platelet count less than 100,000/mm3
8. bilirubin greater than 1.5 mg/dl (> 26 μmol/L, système internationale (SI) unit equivalent)
9. aspartate amino transferase (AST) and/or alanine amino transferase (ALT) greater than 3 times the upper limit of normal
10. serum creatinine greater than 1.5 mg/dl (> 132 μmol/L, SI unit equivalent)
11. concomitant non-oncological diseases which are considered relevant for the evaluation of the safety of the trial drug
12. chemo- or immunotherapy within the past four weeks prior to treatment with the trial drug or during the trial (except for present trial drug)
13. radiotherapy to breast and thorax region within the past four weeks before inclusion or during the trial
14. women who are sexually active and unwilling to use a medically acceptable method of contraception
15. pregnancy or lactation
16. treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial (except for present trial drug)
17. patients unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-10-01 (Actual); Primary Completion 2004-12-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of bivatuzumab mertansine | up to day 21

SECONDARY OUTCOMES:
Incidence of adverse events | up to day 21
Number of patients with clinically significant findings in laboratory tests | up to day 21
Number of patients with clinically significant findings in vital signs | up to day 21
Tumor response rate | up to 1 year
  assessed by response evaluation criteria in solid tumours (RECIST)
Concentration of bivatuzumab mertansine | up to day 21
Concentration of CD44v6 recognising IgG antibodies (anti-CD44v6-IgG) | up to day 21
Number of patients with development of human anti-human antibodies (HAHA) | up to day 21

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency